CLINICAL TRIAL: NCT01061112
Title: Effects of Genotype on CYP2C9 Drug Interactions
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0812M56082; R01GM069753 (NIH)
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: Drug Interactions; Genetics; CYP2C9; Healthy Volunteers
MeSH Terms: interventions — Flurbiprofen; Fluconazole; Ketoprofen; Tolbutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urine samples are to be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CYP2C9*1/*1 Genotype: This genotype is considered the wild type genotype. Individuals with the CYP2C9*1/*1 genotype have two *1 alleles and participated in the following interventions: Flurbiprofen Control - Flurbiprofen Only, Flurbiprofen Inhibition - Flurbiprofen & Fluconazole, Ketoprofen Control - Ketoprofen Only, Ketoprofen Inhibition - Ketoprofen & Fluconazole, Tolbutamide Control - Tolbutamide Only, and Tolbutamide Inhibition - Tolbutamide & Fluconazole.
  Interventions: Drug: Flurbiprofen Control - Flurbiprofen Only; Drug: Flurbiprofen Inhibition - Flurbiprofen & Fluconazole; Drug: Ketoprofen Control - Ketoprofen Only; Drug: Ketoprofen Inhibition - Ketoprofen & Fluconazole; Drug: Tolbutamide Control - Tolbutamide Only; Drug: Tolbutamide Inhibition - Tolbutamide & Fluconazole
- CYP2C9*1/*3 Genotype: Individuals with the CYP2C9*1/*3 genotype have one *1 allele and one *3 allele and participated in the following interventions: Flurbiprofen Control - Flurbiprofen Only, Flurbiprofen Inhibition - Flurbiprofen & Fluconazole, Ketoprofen Control - Ketoprofen Only, Ketoprofen Inhibition - Ketoprofen & Fluconazole, Tolbutamide Control - Tolbutamide Only, and Tolbutamide Inhibition - Tolbutamide & Fluconazole.
  Interventions: Drug: Flurbiprofen Control - Flurbiprofen Only; Drug: Flurbiprofen Inhibition - Flurbiprofen & Fluconazole; Drug: Ketoprofen Control - Ketoprofen Only; Drug: Ketoprofen Inhibition - Ketoprofen & Fluconazole; Drug: Tolbutamide Control - Tolbutamide Only; Drug: Tolbutamide Inhibition - Tolbutamide & Fluconazole
- CYP2C9*3/*3 Genotype: Individuals with the CYP2C9*3/*3 genotype have two *3 alleles and participated in the following interventions: Flurbiprofen Control - Flurbiprofen Only, Flurbiprofen Inhibition - Flurbiprofen & Fluconazole, Ketoprofen Control - Ketoprofen Only, Ketoprofen Inhibition - Ketoprofen & Fluconazole, Tolbutamide Control - Tolbutamide Only, and Tolbutamide Inhibition - Tolbutamide & Fluconazole.
  Interventions: Drug: Flurbiprofen Control - Flurbiprofen Only; Drug: Flurbiprofen Inhibition - Flurbiprofen & Fluconazole; Drug: Ketoprofen Control - Ketoprofen Only; Drug: Ketoprofen Inhibition - Ketoprofen & Fluconazole; Drug: Tolbutamide Control - Tolbutamide Only; Drug: Tolbutamide Inhibition - Tolbutamide & Fluconazole

INTERVENTIONS:
Drug: Flurbiprofen Control - Flurbiprofen Only — A single 50 mg flurbiprofen dose taken at the start of the study period. No other drugs administered during this study period.
  Other Names: Ansaid
Drug: Flurbiprofen Inhibition - Flurbiprofen & Fluconazole — A single 50 mg flurbiprofen dose taken at the start of the study period. 400 mg fluconazole taken every morning starting a week before the start of the study period and continuing throughout the study period.
  Other Names: Ansaid; Diflucan
Drug: Ketoprofen Control - Ketoprofen Only — A single 75 mg ketoprofen dose taken at the start of the study period. No other drugs administered during this study period.
  Other Names: Orudis
Drug: Ketoprofen Inhibition - Ketoprofen & Fluconazole — A single 75 mg ketoprofen dose taken at the start of the study period. 400 mg fluconazole taken every morning starting a week before the start of the study period and continuing throughout the study period.
  Other Names: Orudis; Diflucan
Drug: Tolbutamide Control - Tolbutamide Only — A single 500 mg tolbutamide dose taken at the start of the study period. No other drugs administered during this study period.
  Other Names: Orinase
Drug: Tolbutamide Inhibition - Tolbutamide & Fluconazole — A single 500 mg tolbutamide dose taken at the start of the study period. 400 mg fluconazole taken every morning starting a week before the start of the study period and continuing throughout the study period.
  Other Names: Orinase; Diflucan

SUMMARY:
This research study will help determine how a person's genetic makeup affects their responses to drugs, the ability of the body to break down drugs, and their potential to experience an interaction between drugs. We are investigating the drug interactions between an antifungal drug called fluconazole and the commonly used drugs tolbutamide, flurbiprofen, and ketoprofen. Tolbutamide is used for management of Type 2 diabetes. Both flurbiprofen and ketoprofen are non-steroidal anti-inflammatory drugs (NSAIDs) often used for arthritis or pain. We are interested in studying whether individuals with certain genetic profiles have different drug interactions than normal. This research is being done to see if certain genetic profiles require us to adjust medication doses differently than is needed for the general population. Genetic profiles of subjects are determined from their previous participation in the Pharmacogenetics Registry (Investigator Richard Brundage, University of Minnesota).

The study hypothesis is: Fraction metabolized by CYP2C9 enzyme determines the extent of drug interactions in CYP2C9*1/*1 individuals but this factor (fraction metabolized) becomes less influential and drug interactions are attenuated in a gene-dose dependent manner in individuals with one or more defective alleles.

DETAILED DESCRIPTION:
The study hypothesis is: Fraction metabolized by CYP2C9 enzyme determines the extent of drug interactions in CYP2C9*1/*1 individuals but this factor (fraction metabolized) becomes less influential and drug interactions are attenuated in a gene-dose dependent manner in individuals with one or more defective alleles.

Objective: Examine the extent of fluconazole inhibition of drugs with varying degrees of fraction metabolized by CYP2C9 in individuals with the CYP2C9*1/*1, CYP2C9*1/*3 and CYP2C9*3/*3 genotypes.

People differ in their genetic makeup. This includes differences in genes involved in drug metabolism, transport, and effect in the body. People with certain genetic profiles produce altered enzymes, transporters, and receptors that may respond in different ways to drugs. Altered enzymes cause some drugs to be broken down at a different rate than normal. As a result, drug concentrations build up in the blood, and increase the risk of side effects. Furthermore, when two drugs are taken together, the possibility exists for the drugs to interact, with one drug causing a change in the metabolism of the other or both of the drugs. It is not known whether people with an altered genetic makeup also have an altered experience with drug interactions. Altered drug transporters can affect the absorption and elimination of drugs as compared to normal causing differences in how long the drug stays in the body. Finally, altered drug receptors can respond differently to drugs and, thus, produce altered desired or undesired effects.

In this study, we will be investigating the drug interactions between an antifungal drug called fluconazole and the commonly used drugs tolbutamide, flurbiprofen, and ketoprofen in subjects with three different genotypes of the CYP2C9 enzyme. Tolbutamide is used for management of Type 2 diabetes. Both flurbiprofen and ketoprofen are non-steroidal anti-inflammatory drugs (NSAIDs) often used for arthritis or pain. We are interested in studying whether individuals with certain genetic profiles have different drug interactions than normal. This research is being done to see if certain genetic profiles require us to adjust medication doses differently than is needed for the general population.

The cytochrome P450 (CYP) superfamily of enzymes plays an important role in the oxidative conversion of numerous xenobiotics into their more hydrophilic metabolites. CYP2C9, is an important member of the CYP superfamily, accounting for 10-20% of the CYP protein content in human liver and catalyzes approximately 20% of the CYP mediated drug oxidation reactions, including tolbutamide and the non-steroidal anti-inflammatory drugs (NSAIDs) such as ketoprofen and flurbiprofen. It is now well established that genetic factors play an important role in the control of CYP2C9 expression and activity. In particular, the *3 allele is expressed at an allele frequency of 15%. Homozygotic *3 individuals exhibit significantly reduced oral clearance for several CYP2C9 substrates. In most of these cases, the reduction in clearance approaches 80% and even in heterozygotic individuals, this reduction in clearance is 40-50% due to the co-dominant expression of CYP2C9. This reduction in clearance has been associated with an increased frequency of adverse events following warfarin or phenytoin administration, two clinically important drugs that exhibit a narrow therapeutic index. The therapeutic index is a comparison of the amount of a therapeutic agent that causes the therapeutic effect to the amount that causes toxic effects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be 18-60 years old.
* Women of child-bearing age must be willing to use measures to avoid conception during the study period.
* Subjects must agree not to take any known substrates, inhibitors, inducers, or activators of CYP2C9.

Exclusion Criteria:

* Current cigarette smoker.
* Abnormal renal or liver function tests, physical exam, or recent history of hepatic, renal, gastrointestinal or neoplastic disease.
* Allergy to tolbutamide, flurbiprofen, ketoprofen, fluconazole or phenytoin and other chemically related drugs.
* Recent ingestion (< 1 week) of any medication known to be metabolized by or alter activity of CYP2C9.
* A positive pregnancy test during the time of the pharmacokinetic study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects are selected from a pharmacogenetics registry in which their drug metabolism genotype has been determined.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Flurbiprofen Clearance | 48 hours post Flurbiprofen dose
  Measure of blood concentrations of Flurbiprofen 48 hours post Flurbiprofen dose
Ketoprofen Clearance | 48 hours post Ketoprofen dose
  Measure of blood concentrations of Ketoprofen 48 hours post Ketoprofen dose
Tolbutamide Clearance | 48 hours post Tolbutamide dose
  Measure of blood concentrations of Tolbutamide 48 hours post Tolbutamide dose

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brundage, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Clinical and Translational Science Institute, Minneapolis, Minnesota, United States